CLINICAL TRIAL: NCT00826826
Title: The Effect of Short Term Amiodarone Treatment on Success Rate and Quality of Life After Catheter Ablation for Atrial Fibrillation
Brief Title: The Effect of Short Term Amiodarone Treatment After Catheter Ablation for Atrial Fibrillation
Acronym: AMIO-CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Stine Darkner, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-A-2008-085; H-A-2008-085; 2612-3819; 2008-004500-32
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Amiodarone; Arrhythmias, Cardiac; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Catheter Ablation; Amiodarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amiodarone (Active Comparator)
  Interventions: Procedure: Catheter ablation; Drug: Amiodarone
- Placebo (Placebo Comparator)
  Interventions: Procedure: Catheter ablation; Drug: Placebo

INTERVENTIONS:
Procedure: Catheter ablation — (Pulmonary vein isolation)
Drug: Amiodarone — From the day of the catheter ablation procedure and 8 weeks forward.
  Arms: Amiodarone
Drug: Placebo — From the day of the catheter ablation procedure and 8 weeks forward.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the overall effectiveness of short-time anti-arrhythmic drug treatment with amiodarone (to control heart rhythm) to prevent short-and long-term atrial fibrillation following an ablation procedure for atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia, and it is associated with increased mortality and morbidity due to increased risk of stroke, poor quality of life and risk of developing heart failure.

Today, catheter ablation has become a standard procedure in the treatment of symptomatic atrial fibrillation, but so far there is no official recommendations regarding the use of antiarrythmic drugs after the procedure. Nevertheless, it is common standard practice to prescribe antiarrhythmic drugs for the first 2-3 months after the intervention to prevent early recurrences. To our knowledge, the effect of antiarrythmic drugs following ablation for atrial fibrillation has only been evaluated in a few recent studies. None of these have evaluated the long term effect of short term antiarrythmic drug treatment. In addition, none of the trials have been conducted placebo-controlled.

In this study patients with paroxysmal or persistent atrial fibrillation will be considered for randomisation. Following the ablation procedure, patients will be randomized to receive either amiodarone or placebo for a period of 8 weeks. Clinical visits including a physical exam, 12 lead ECG recording and blood samples, will be scheduled during the follow-up time. Furthermore patients will be evaluated with Quality of Life questionaires and Holter monitoring.

The primary endpoint of the study is freedom from atrial fibrillation, atrial flutter or atrial tachycardia at 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic paroxysmal or persistent atrial fibrillation undergoing catheter ablation for atrial fibrillation. (persistent episodes may last no more than 12 months)

Exclusion Criteria:

* Contraindication or intolerance to amiodarone.
* Prolonged amiodarone treatment within 3 months before the planned ablation procedure.
* Previous participation in this study.
* Other cardiac arrythmias (patients with co-existing atrial flutter can be included).
* Antiarrhythmic treatment for indication other than atrial fibrillation (or atrial flutter).
* Heart failure (NYHA class III or IV or left ventricular ejection fraction < 35%).
* Significant heart valve disease.
* Significant lung disease, thyroid dysfunction or liver disease.
* Inability or unwillingness to be treated with anticoagulation before and during the study.
* Females with birth giving potential
* Failure to give informed concent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2009-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation, atrial flutter or atrial tachycardia. | 6 months from ablation procedure
  Patients who (based upon clinical decision) are re-ablated within the blanking period counts as having reached an end point.

SECONDARY OUTCOMES:
Quality of Life | 6 months
Adverse outcome/intolerance of antiarrhythmic agent requiring cessation of drug | 6 months
Structural and electrical changes (evaluated by echocardiography and digital ECG). | 6 months
Atrial fibrillation burden evaluated by Holter monitoring | 6 months
Asymptomatic atrial fibrillation, atrial flutter or atrial tachycardia documented with Holter. | 6 months
Within blanking period of 3 months: Number AF-related hospitalisations, need for cardioversion or need for additional antiarrythmic drugs. | 3 months
Symptom burden. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stine Darkner, MD, Principal Investigator — Rigshospitalet, Denmark; Jesper H Svendsen, MD, DMSc, Study Director — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Gentofte University Hospital, Hellerup

REFERENCES:
- [Derived] Olsen FJ, Darkner S, Chen X, Pehrson S, Johannessen A, Hansen J, Svendsen JH, Biering-Sorensen T. Effect of Amiodarone after Catheter Ablation According to Left Atrial Structure and Function: The AMIO-CAT Trial. Am J Cardiol. 2026 Jan 15;259:63-70. doi: 10.1016/j.amjcard.2025.09.017. Epub 2025 Sep 24. PMID 41005596